CLINICAL TRIAL: NCT04205383
Title: Quantification of the Main Circulating Histones During Normal Pregnancy and Pregnancies With Placenta-mediated Complications
Brief Title: GROSS-HIST : Quantification of the Main Circulating Histones During Normal Pregnancy and Pregnancies With Placenta-mediated Complications
Acronym: GROSS-HIST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Nimao/2018-03/SB-01
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy; Pregnancy Complications; Healthy Volunteers
MeSH Terms: conditions — Pregnancy Complications | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pregnancy: pregnant women with normal pregnancy
  Interventions: Other: biological analyses
- pregnancy with complications: pregnant women with placental-mediated complications of pregnancy type complications
  Interventions: Other: biological analyses
- healthy volunteer: healthy, non-pregnant women volunteers
  Interventions: Other: biological analyses

INTERVENTIONS:
Other: biological analyses — The histones H3-citrullinated, acetylated histones (Pan-histones), H1 histone as well as the free HMGB1 protein will be quantified. This choice corresponds to the histones involved in inflammation, proliferation, migration or cell differentiation and can be quantified to date.

SUMMARY:
Pregnancy generates an increased thrombotic risk, and placental-mediated diseases are a risk factor for cardiovascular diseases, in particular: pre-eclampsia (PE), intrauterine growth retardation (IUGR), retroplacental hematomas (HRP), late intrauterine fetal deaths (LIFD) of placental origin and preterm deliveries of vascular origin. They are responsible for significant maternal-fetal morbidity/mortality. Data published in 2007 by the Haute Autorité de Santé (HAS) show that hypertension and pre-eclampsia are, in France, at the origin of 3 to 8% of the risk of perinatal mortality.

During pregnancy, a transitional organ of foetal origin, the placenta, is established, which is essential for the maintenance and harmonious development of the pregnancy. The chorionic villus, in contact with maternal blood in the intervillous chamber, is the structural and functional unit of the placenta. After the initial implantation phase, the trophoblastic cell constituting the main part of the placental villi differs in two ways: (A) into "citrus cytotrophoblasts" whose cells will fuse to generate the multinucleated outer layer giving the syncytiotrophoblast that ensures fetal-maternal exchanges and endocrine functions of the placenta; (B) into "invasive extra-city cytotrophoblasts" essential for the effective anchoring of the placenta in the decidualized uterine mucosa and for the remodelling of the terminal uterine spiral arteries, whose resistance to blood flow must collapse to allow effective oxygenation of the villi. Extra-city trophoblasts change from an epithelial phenotype to an endothelial phenotype. They may thus be exposed to pro-thrombotic factors such as endothelial cells. A lack of trophoblastic invasion and incomplete remodelling of the spiral uterine arteries are responsible for placental hypo-perfusion, hypoxia and the occurrence of placenta-mediated pathologies (pre-eclampsia, intrauterine growth retardation, retroplacental hematoma, fetal loss and fetal death in utero). The most common placental-mediated disease is pre-eclampsia (5% of births). It corresponds to a complication occurring from the second trimester of pregnancy and which is clinically characterized by high blood pressure, oedema and proteinuria. It is responsible for premature deliveries and is a major cause of intrauterine growth restriction.

To date, there is no specific and early biomarker for the occurrence of placental vascular pathologies. Recent developments raise, for example, the question of circulating angiogenesis inhibitory factors (sFlt1, sEng) in pre-eclampsia. With regard to treatment, early administration of low-dose aspirin before 16 weeks of pregnancy seems to reduce the risk of pre-eclampsia, hence the importance of having very early markers of the disease. Discovering such markers is therefore one of the major challenges in strengthening women's follow-up and avoiding subsequent complications. For fetal losses and retroplacental hematoma, the administration of low molecular weight heparin has been shown to be effective. However, these treatments are not specific to placental vascular pathologies. Thus, understanding and exploring the cellular and molecular mechanisms of vascular-placental interface dysfunctions remains necessary to enable targeted management of patients feeding the general principle of precision medicine.

Compare the concentrations of (i) circulating histones involved in inflammation, proliferation, migration or cell differentiation (H3-citrullinated histone, acetylated histones (Pan-histones), H1 histone) and (ii) free HMGB1 protein between the three patient groups ("GrossN", "GrossC", "VolS").

The histones H3-citrullinated, acetylated histones (Pan-histones), H1 histone as well as the free HMGB1 protein will be quantified. This choice corresponds to the histones involved in inflammation, proliferation, migration or cell differentiation and can be quantified to date.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria :
* The patient must have given her free and informed consent and signed the consent
* The patient must be a member or beneficiary of a health insurance plan
* Only women are included
* The patient is at least 18 years old
* Inclusion criteria for the target population:
* pregnant patient with a complication of the placental vascular pathology type (pre-eclampsia, eclampsia, HELLP syndrome, retroplacental hematoma, fetal death in utero) or venous thromboembolic disease (deep vein thrombosis, pulmonary embolism).

OR pregnant woman, without complications (normal pregnancy), absence of identified chronic pathology, absence of a history of neoplastic pathology, absence of a history of thromboembolic disease, absence of a history of chronic infectious pathology, absence of acute pathology (benign infectious type) intercurrent within the previous 2 weeks.

OR

- female, healthy volunteer, non-pregnant, no identified chronic pathology, no history of neoplastic pathology, no history of thromboembolic disease, no history of chronic infectious pathology, no history of acute (benign infectious type) intercurrent pathology within the previous 2 weeks.

Exclusion Criteria:

* General non-inclusion criteria :
* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under the protection of justice, under guardianship or curatorship
* Patient refuses to sign consent
* It is impossible to give informed information about
* The patient does not read French fluently

Criteria for non-inclusion regarding interfering diseases or associated conditions:

* The patient is undergoing hormonal ovarian stimulation treatment as part of medically assisted reproduction
* The patient is pregnant OR
* The patient is breastfeeding OR
* The patient has been giving birth for less than 3 months .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant patient with a complication of the placental vascular pathology type (pre-eclampsia, eclampsia, HELLP syndrome, retroplacental hematoma, fetal death in utero) or venous thromboembolic disease (deep vein thrombosis, pulmonary embolism).
  AND pregnant woman, without complications (normal pregnancy), absence of identified chronic pathology, absence of a history of neoplastic pathology, absence of a history of thromboembolic disease, absence of a history of chronic infectious pathology, absence of acute pathology (benign infectious type) intercurrent within the previous 2 weeks.
  AND
  - female, healthy volunteer, non-pregnant, no identified chronic pathology, no history of neoplastic pathology, no history of thromboembolic disease, no history of chronic infectious pathology, no history of acute (benign infectious type) intercurrent pathology within the previous 2 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Circulating levels : Protein HMGB1 ng/ml | until the patient gives birth, up to 7 months on average
  Protein HMGB1 ng/ml
Circulating levels : Citrullinated Histone H3 U/ml | until the patient gives birth, up to 7 months on average
  Citrullined Histone H3 U/ml
Circulating levels : Histone H1 U/ml | until the patient gives birth, up to 7 months on average
  Histone H1 U/ml
Circulating levels : Acetylated Histones U/ml | until the patient gives birth, up to 7 months on average
  Acetylated Histones U/ml
Circulating levels : Histone H3 U/ml | until the patient gives birth, up to 7 months on average
  Histone H3 U/ml

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bouvier S, Fortier M, Vincent L, Demattei C, Mousty E, Herzog M, Rommelaere G, Nouvellon E, Mercier E, Letouzey V, Gris JC. NETosis Markers in Pregnancy: Effects Differ According to Histone Subtypes. Thromb Haemost. 2021 Jul;121(7):877-890. doi: 10.1055/s-0040-1722225. Epub 2021 Jan 10. PMID 33423243